CLINICAL TRIAL: NCT04527224
Title: A Phase I/Ⅱa Trial to Explore the Safety and Efficacy of Allogenic Adipose Tissue-derived Mesenchymal Stem Cell (AstroStem-V) Therapy in Patients With COVID-19 Pneumonia
Brief Title: Study to Evaluate the Efficacy and Safety of AstroStem-V in Treatment of COVID-19 Pneumonia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nature Cell Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASVP1N2A-US
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Covid19 Pneumonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AstroStem-V (Experimental): AstroStem-V which consists of three syringes and each syringe contains 1.0 x 10^8 cells / 3mL of saline with 30% human serum
  Interventions: Drug: AstroStem-V

INTERVENTIONS:
Drug: AstroStem-V — Allogenic adipose tissue-derived mesenchymal stem cells (AdMSCs)

SUMMARY:
This study is an open-label, single-arm study to evaluate the safety and efficacy of Astrostem-V, allogenic adipose tissue derived mesenchymal stem cells (AdMSC), in patients with COVID-19 pneumonia. After each subject completes 12-Weeks visit (Visit 12) and the data management team confirms all individual data have no issue, the individual database will be locked and the blinding will be open for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 80 years at the time of signing the written consent form
* Subjects diagnosed with pneumonia by radiologic examination (Chest X-ray or CT) at screening and baseline
* subject who has moderate COVID-19 disease:

  * Subjects have laboratory-confirmed SARS-CoV-2 infection within 28 days from screening by authorized a reverse-transcription polymerase chain reaction (RT-PCR) or equivalent testing at baseline
  * A subject who has symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion
  * A subject who has clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≤ 20 breaths per minute, SpO2 ≥ 93% on room air at sea level, heart rate ≤ 90 beats per minute
  * No clinical signs indicative of severe COVID-19 disease severity
* Subjects voluntarily participate in the clinical trial with written informed consent

Exclusion Criteria:

* Subjects who have pulmonary disease except COVID-19 pneumonia
* SpO2 ≤ 93%
* Subjects who have uncontrolled shock
* Subjects diagnosed with COVID-19 with CPR or requires treatment of Extra Corporeal Membrane Oxygenation (ECMO)
* Subjects with an irreversible brain lesion or medical history of malignant tumors
* Subjects treated for heart disease within 3 months prior to screening
* Subjects who are receiving immunosuppressant therapy for transplantation or who are taking immunosuppressive drugs such as steroids, TNF-alpha inhibitors
* Subject treated with stem cells.
* Subjects with end-stage renal failure who need renal replacement therapy or cirrhosis patients with complications
* Subjects who have an average life expectancy to be less than 2 months due to the underlying disease
* Subjects who have history of thromboembolism or pulmonary arterial hypertension
* Subjects who currently have positive HIV test results
* Pregnant or breast-feeding women
* Subjects with pregnancy planned during clinical trials. Women or men of childbearing age who do not agree to maintain contraception by choosing, or who do not agree to use the appropriate method of contraception

  * suitable contraceptive methods: condom, sponge, foam, gel, diaphragm for contraception, intrauterine device, etc. Periodic abstinence (eg, calendar method, ovulation method, symptom body temperature method, post ovulation method) and restraint is not considered an accepted method of contraception, and hormonal contraceptives are not allowed. However, women having no potential are pregnancy due to menopause (amenorrhea more than 12 months after the last menstruation) or surgical infertility is possible to participate in the study only the pregnancy test is negative
* Subjects who administered other investigational products within 12 weeks prior to IP administration
* Subject who the principal investigator considers inappropriate for the study due to any other reasons than those listed above
* Subjects who cannot tolerate aspirin

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From baseline to Week 12
  Number of subjects with treatment related adverse events as assessed by analysis of adverse events including symptoms.
Abnormalities of physical examination, vital signs, and laboratory test | From baseline to Week 12
  Number of subjects with treatment related adverse events as assessed by analysis of adverse events including abnormal findings on physical examination, vital signs, ECG, and standard laboratory examination.

SECONDARY OUTCOMES:
SpO2 | From baseline to Week 12
  Change from baseline in SpO2 at every visit
Mortality rate | Week 4, Week 8, and Week 12
  Check survival status of the subject at Visit 6, 10(Week 4, 8 and Week 12 if follow-up is possible) and record the status on eCRF.
Ventilator treatment status | From Week 1 to Week 12
  Check the duration of the ventilator retention, check when the ventilator treatment has been completed after the baseline.
Improvement of pneumonia assessed by radiologic examination(Chest X-ray or CT) | From baseline to Week 12
  Perform chest X-ray every week (W1-W12) after screening, baseline, and W1 followed by 2-week intervals (W1, W2, W4, W6, W8, W12). In addition, CT is measured at week baseline, W4, W8 and W12.
SOFA score (Sequential Organ Failure Assessment) | From baseline to Week 12
  Check the SOFA score every week (W1-W12) after baseline, and W1 followed by 2-week intervals (W1, W2, W4, W6, W8, W12).
  Choose the worst of the six physiological measurements and score between 0 and 4 points each and check the total. If the measured value is more than 3 points, it is defined as organ failure.
2019 nCOV nucleic acid test | From baseline to Week 12
  The Real-time PCR (RT-PCR) test for COVID-19 is measured at 2-week intervals (W1-W12) from Screening, Baseline to W1, W2, W4, W6, W8 and W12.

CONTACTS AND LOCATIONS:
Overall Officials: JeongChan Ra, Ph.D., Study Director — Nature Cell Co. Ltd.
Locations (2):
- United States (2):
  - Medical Advancement Center of Arizona, Phoenix, Arizona
  - Epic Medical Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided